CLINICAL TRIAL: NCT00904553
Title: Pilot Study of Resection Combined With Stereotactic Radiosurgery in Patients With Limited (1-3) Brain Metastases
Brief Title: Study of Resection Combined With Stereotactic Radiosurgery for 1 to 3 Brain Metastases
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Michael Milano, MD,PhD, Associate Professor, University of Rochester
Other Study IDs: URBT07099; RSRB00023405 (Other: Univ of Rochester IRB)
Record Dates: First submitted 2009-05-15; First posted 2009-05-19 (Estimated); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Neoplasm Metastasis
Keywords: Brain; metastases
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — brain tissue
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Novalis Shaped Beam Surgery: Patients with limited brain metastases (mostly solitary brain metastasis) treated with Novalis Shaped Beam Surgery followed by planned craniotomy and resection of the metastases.
  Interventions: Radiation: Novalis Shaped Beam Surgery

INTERVENTIONS:
Radiation: Novalis Shaped Beam Surgery — Treatment using Novalis SRS

SUMMARY:
This study is to look more closely at the tumor removed during your surgery, and to follow your condition after your treatment.

The purpose of this study is to determine what side effects are common or more rare from this treatment, how well the treatment has worked for you, and to track whether you develop other brain metastases.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a previously histopathologically proven diagnosis of malignancy.
* Patients must be evaluated by Neurosurgery and Radiation Oncology
* Patients must have 1-3 brain metastases seen on MRI or CT imaging. At least one brain metastases must be considered resectable by craniotomy as determined by the treating neurosurgeon. Brain lesion resection must be considered standard of care. A not uncommon situation is for a patient to undergo resection of a solitary metastasis, but prove to have more lesions on subsequent MRIs (perhaps too small to be seen on a pre-operative MRI). These patients will be eligible if the total number of lesions is 1-3.
* All lesions must be treatable by SRS as determined by the treating neurosurgeon and radiation oncologist.
* All lesions must be <4 cm in greatest dimension. For patients with more than 1 brain metastases, only 1 lesion can exceed 3 cm in greatest dimension.
* In patients treated to the post-op surgical cavity, this cavity must be encompassed by a CTV of <5 cm.
* Patients must have a Karnofsky performance status ≥60.
* Extracranial disease must not be considered imminently life threatening (<2 month anticipated survival from extracranial disease).
* Patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines.

Exclusion Criteria:

* KPS<60
* life expectancy > 2 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated at the University of Rochester Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2009-01-14 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2022-03-28 (Actual)

PRIMARY OUTCOMES:
Determine toxicity of treatment with cranial SRS and resection | During treatment and long term follow-up
Determine the local control of the treated lesion(s), distant brain control and overall patient survival. | During treatment and long term follow-up

SECONDARY OUTCOMES:
Tissue from the resected brain metastases will be evaluated with immunohistochemistry and/or comparative genomic hybridization to assess for potential markers for clinical outcome as well as potential markers of radiation response. | Following surgical resection

CONTACTS AND LOCATIONS:
Overall Officials: Michael Milano, MD PhD, Principal Investigator — Department of Radiation Oncology, University of Rochester Medical Center
Locations (1):
- Department of Radiation Oncology, University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No